CLINICAL TRIAL: NCT04883762
Title: Fecal Microbiota Transplantation (FMT) for Immune Checkpoint Inhibitor (ICI)-Related Diarrhea: A Pilot Study
Brief Title: Stool Transplant to Control Treatment-related Diarrhea
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-242
Record Dates: First submitted 2021-05-10; First posted 2021-05-12 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Fecal Microbiota Transplantation (FMT)
Keywords: Immune Checkpoint Inhibitor (ICI)-Related Diarrhea; 20-242
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized pilot trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (FMT) (Experimental): Study subjects will undergo standard bowel preparation and diagnostic colonoscopy with routine biopsies for pathologic assessment. FMT will be performed at the proximal extent of the colon reached, according to the same protocol used in prior randomized studies. FMT will use healthy donor stool provided by OpenBiome, a nonprofit 501(c)(3) organization that provides clinicians and hospitals with screened, filtered and frozen stool to be used for FMT. Routine clinical and research biopsies will be collected during the FMT colonoscopy procedure.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — Undergo FMT via colonoscopy.

SUMMARY:
This study will test the safety, effectiveness, and feasibility of a treatment called fecal microbiota transplantation (FMT) to reduce the symptoms of ICI-related diarrhea.

FMT uses a liquid preparation of stool collected from a healthy donor with normal (healthy) bacteria; this liquid is infused into the small or large intestine of a recipient during a colonoscopy procedure. The study researchers think that the healthy bacteria in the transplanted stool will grow and replace the unhealthy bacteria and return the intestines and colon of the recipient to a healthy state.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Patient has been treated with immune checkpoint inhibitors (ICI), including anti-CTLA-4, anti-PD-1 and anti-PDL-1 therapy for any malignant indication
* Patient has developed diarrhea ≥ Grade 2 attributed to ICI
* Patient has diarrhea ≥ Grade 2 attributed to ICI, that persists despite treatment with corticosteroids for at least 72 hours and/or at least one dose of a biologic medication, such as infliximab or vedolizumab, with symptoms that persist or recur at least 72 hours post-infusion ° If no to the above, patient has a contraindictation to immunosuppressive treatment

Exclusion Criteria:

* Active GI infection, including untreated viral, bacterial or fungal or alternative identified cause(s) of diarrhea.
* Antibiotic exposure within 48 hours prior to FMT
* Expected prolonged compromised immunity indicated by at least one of the below:

  * Known HIV infection with CD4 count <240
  * ANC <1000/mm3 (use of growth factors to raise ANC is acceptable)
* Seronegative for EBV or CMV (i.e. EBV IgG negative or CMV IgG negative)
* Contraindications to anesthesia for procedure indicated by at least one of the below:

  * Serious cardiopulmonary comorbidities
  * Inability to tolerate anesthesia
* Pregnancy

  * Patient is pregnant
  * Women of childbearing potential should not have plans to became pregnant or breastfeed an infant and must agree to use a highly effective method of birth control until 2 months after treatment with FMT (e.g. barrier method, oral or parenteral contraceptives, a vasectomized partner, or abstinence from sexual intercourse)
* Severe food allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of fecal microbiota transplantation (FMT)-related adverse events | for 7 days after each FMT
  will be grading according to CTCAE 5.0.1

CONTACTS AND LOCATIONS:
Overall Officials: David Faleck, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm